CLINICAL TRIAL: NCT04363125
Title: Systematic Review of Isolated Hypoganglionosis and Presentation of a New Case Complicated With Sigmoid Volvulus
Brief Title: Review of Isolated Hypoganglionosis and Presentation of a New Case Complicated With Sigmoid Volvulus
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Ufuk Uylas, Principal Investigator, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: 23042020
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Pathology; Sigmoid Volvulus; Hypoganglionosis
Keywords: colon; constipation; derotation; obstruction; Hypoganglionosis; intestinal neuronal dysplasia
MeSH Terms: conditions — Constipation; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pathology result — Pathology result of rectal biopsy

SUMMARY:
Isolated hypoganglionosis is rare and constitutes 3-5% of all congenital neurological bowel diseases. Since hypoganglionosis is associated with symptoms such as chronic constipation or pseudo-obstruction, it can be confused with Hirschprung's disease and it is important to make a differential diagnosis before treatment. Our aim in this study; In addition to sharing the rarely isolated hypoganglionosis and sigmoid volvulus in a 45-year-old male patient with mental retardation, the investigators present a systematic comprehensive review of hypoganglionosis.

DETAILED DESCRIPTION:
Isolated hypoganglionosis is rare and constitutes 3-5% of all congenital neurological bowel diseases. Since hypoganglionosis is associated with symptoms such as chronic constipation or pseudo-obstruction, it can be confused with Hirschprung's disease and it is important to make a differential diagnosis before treatment. Our aim in this study; In addition to sharing the rarely isolated hypoganglionosis and sigmoid volvulus in a 45-year-old male patient with mental retardation, the investigators present a systematic comprehensive review of hypoganglionosis. Pubmed and Scopus databases were scanned. No restrictions were used in the written language. Only isolated cases of hypoganglionosis were added to the study. In the cases; author, year of publication, country of publication, age, gender, surgical or non-surgical treatments, treatment results, and mortalities were examined.

When sigmoid volvulus is seen in children and adolescents, congenital neurological bowel diseases should be considered in the differential diagnosis. Hirschprung's disease must be ruled out by rectal biopsy. The histopathological investigation should be carried out for the diagnosis and determination of surgical margins in isolated hypoganglionosis.

ELIGIBILITY:
Inclusion Criteria:

* isolated hypoganglionosis
* our case of isolated hypoganglionosis

Exclusion Criteria:

* hypoganglionosis with Hirschsprung's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: our case of isolated hypoganglionosis and published isolated hypoganglionosis studies patients.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Mortality | three months
  Mortality of sigmoid volvulus due to isolated hypoganglionosis

CONTACTS AND LOCATIONS:
Overall Officials: ufuk uylas, Specialist, Principal Investigator — Dr. Ersin Arslan Training and Resource Hospital
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)